CLINICAL TRIAL: NCT02099695
Title: Clinical Trial Phase III, Prospective, Randomized, Double-blind, Multicenter, National, Comparative Between Oxybutynin Chloride With Placebo to Evaluate the Efficacy and Safety for Systemic Treatment of Primary Hyperhidrosis.
Brief Title: Evaluate the Efficacy of Oxybutynin Chloride in Patients With Primary Hyperhidrosis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The company changed the strategy.
Sponsor: Cristália Produtos Químicos Farmacêuticos Ltda. (Industry)
Collaborators: Hospital Israelita Albert Einstein (Other); University of Sao Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRT069
Record Dates: First submitted 2014-03-20; First posted 2014-03-31 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Hyperhidrosis
Keywords: Hyperhidrosis; Oxybutynin
MeSH Terms: conditions — Hyperhidrosis | interventions — oxybutynin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxybutynin Chloride (Active Comparator): * Tablet
  * Dose 5,0 or 10 mg/ day
  Interventions: Drug: Oxybutynin
- Placebo (Placebo Comparator): - Tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxybutynin — The doses will increase due to the absence/ lack of therapeutic response of the previous dose assessed during the study visits.
  Arms: Oxybutynin Chloride
Drug: Placebo — The quantity of tablets will increase due to the absence/ lack of therapeutic response.
  Arms: Placebo

SUMMARY:
Treatment of primary hyperhidrosis through a comparative study between oxybutynin hydrochloride and placebo.

Hydrochloride may decrease the symptoms of hyperhidrosis improving the subject's quality of life.

DETAILED DESCRIPTION:
Clinical Trial phase III, randomized, national, prospective, double-blind, multicenter, comparative between oxybutynin hydrochloride and placebo, to be held in participants aged over 18 years to evaluate the therapeutic efficacy and safety of oxybutynin chloride to systemic treatment of primary hyperhidrosis.

Primary hyperhidrosis is a relatively common disorder, affecting approximately 3% of the population. It affects both sexes similarly and in all age groups, varying only the starting age of symptoms according to the most affected part of the body:

childhood - plantar and palmar hyperhidrosis adolescence - axillary hyperhidrosis adult - craniofacial hyperhidrosis

There is a family history associated with between 12.5% and 56.5% of the participants, according to epidemiological studies.

Initially the subjects will be evaluated on the inclusion and exclusion criteria through screening and safety tests such as blood tests , ECG and tonometry, to confirm enrollment.

When included will be randomized into the corresponding study arm to start study treatment.

During the period of the study it will evaluate the efficacy parameters of the drug.

The treatment for each subject will be about 8 weeks. The inclusion period is foreseen for 6 months and may be extended or decreased according to the pace of inclusion.

The data are summarized according to the study group (per dose and per visit, if applicable) through appropriate descriptive statistics to the variable type. Frequency and percentage will be used for the variables.

The Adverse Events (AE) will be analyzed based on questioning by the investigators in relation to the AE experienced by the subjects. The orientation will be to the subject to note the symptom, the date and time that the event appeared.

ELIGIBILITY:
Inclusion Criteria:

* Understanding, agreement and consent form signed;
* Literate;
* Confirmed diagnosis for primary hyperhidrosis;
* Screening tests at normal standards;
* Absence of pregnancy by Beta-human chorionic gonadotropin test;

Exclusion Criteria:

* Secondary Hyperhidrosis;
* Myasthenia gravis;
* Lactation;
* Hypersensitivity to oxybutynin;
* Use more than 500mg of caffeine;
* Alcoholism;
* Use of illicit drug;
* Changes in ECG (echocardiogram) or tonometry;
* Any clinical condition that the investigator considers clinically significant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2016-01 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Oxybutynin Chloride efficacy | 6 weeks
  Evaluation of the therapeutic efficacy by Oxybutynin Hydrochloride in the treatment of primary hyperhidrosis.

SECONDARY OUTCOMES:
Perception of improvement | During treatment until week 8
  Evaluation of perception of improvement from the subject by completing a questionaire
Evaluate therapeutic safety | During treatment until week 8
  Evaluate therapeutic safety of the Oxybutynin Chloride by assessing possible adverse event
Quality of life | During treatment until week 8
  Evaluate the difference in subject's quality of life between the treatment groups
Time of subject response | End of 8 weeks
  Evaluation of average time the subject reaches response
Duration of response | End of 8 weeks
  Evaluate the duration of response
Evaluation between quality of life and groups | End of 8 weeks
  Evaluate the difference of quality of life in the end of treatment between the groups

CONTACTS AND LOCATIONS:
Overall Officials: José R Milanez de Campos, Principal Investigator — Hospital Israelita Albert Einstein
Locations (2):
- Brazil (2):
  - Hospital Israelita Albert Einstein, São Paulo, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo